CLINICAL TRIAL: NCT06447051
Title: Efficacy of New Post Kasai ILBS Protocol in BiliaryAtresia.
Brief Title: Efficacy of New Post Kasai ILBS Protocol in Biliary Atresia.
Status: Recruiting | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-Biliary Atresia-01
Record Dates: First submitted 2024-06-03; First posted 2024-06-06 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-03

CONDITIONS: Biliary Atresia
MeSH Terms: conditions — Biliary Atresia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Biliary Atresia: Subject undergoing Kasai Surgery at Institute of Liver and Biliary Sciences would be enrolled and will include retrospective historical cohort (Jan 2015 to Dec 2017) and retrospective + prospective cohort with new protocol (Jan 2018 till June 2024).
  Interventions: Other: Kasai Surgery

INTERVENTIONS:
Other: Kasai Surgery — As per institute treatment protocol

SUMMARY:
Biliary atresia (BA) is a neonatal progressive fibrosing cholan- giopathy and the most frequent indication for pediatric liver trans- plantation [1]. Surgical removal of biliary remnants and Roux-en-Y hepatoportoenterostomy (HPE) aims to restore biliary drainage and suppress progression to cirrhosis. Successful HPE, defined as a serum total bilirubin level <2 mg/dL at three months after surgery, occurs in ∼50% of patients in the United States [2]. Young age seems to be the best predictor of response to HPE, with limited data on the efficacy of adjuvant therapies such as corticosteroids, antibiotics, and choleretic agents [3,4]. Potential modes of action of these therapies are to increase bile flow as well as exert an anti- inflammatory effect [5].

In 2007, a double-blind randomized trial in the United Kingdom identified a beneficial effect on corticosteroid therapy on reduction of bilirubin level at one month post HPE without sig- nificant change in the need for liver transplantation [6]. Since then there have been multiple trial most prominent being, Kings hospital trial [7] and START trial [8] which demonstrated reduction in bilirubin levels; however both failed to demonstrate any effect on native liver survival.

However one study done by Bezerra et al [9] where they employed steroid in customised manner showed significant improvement in bile drainage in their subjects versus their historical cohort. Hence we propose to perform a prospective cohort study to assess the Efficacy of new post Kasai (steroid) ILBS protocol in Biliary Atresia.

DETAILED DESCRIPTION:
Study population : Subject undergoing Kasai Sx at Institute of Liver and Biliary Sciences would be enrolled and will include retrospective historical cohort (Jan 2015 to Dec 2017) and retrospective + prospective cohort with new protocol (Jan 2018 till June 2024).

Study design: Cohort study with historical control ( Jan 2015- Dec 2017) Sample size: Time bound. All cases presenting during the study period will be included in the study.

Monitoring and assessment: Liver function test, Hemogram and International Normalised Ratio (INR) would be done weekly for one month, twice weekly for 2nd month and monthly thereafter till 1 year.

Statistical Analysis: Appropriate statistical test for correlation analysis will be applied.

Adverse effects: As per previous studies done , no serious adverse effect has been noted in treatment group vs control group.

ELIGIBILITY:
Inclusion Criteria:

1. Post Kasai Biliary atresia operated at ILBS with retrospective historical cohort (Jan 2015 to Dec 2017) and retrospective + prospective cohort with new protocol (Jan 2018 till June 2024).

Exclusion Criteria:

1. Subjects having major surgical complications
2. Defaulters or Patient not following protocol/not giving consent
3. Biliary atresia splenic malformation

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subject undergoing Kasai Sx at Institute of Liver and Biliary Sciences would be enrolled and will include retrospective historical cohort (Jan 2015 to Dec 2017) and retrospective + prospective cohort with new protocol (Jan 2018 till June 2024).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
We expect steroids used in customized manner to improve biliary drainage and thereby improve native liver survival in post kasai patients. | Within 6 months

SECONDARY OUTCOMES:
Improved survival with native liver at 12 months of age. | 12 months
Reduced progression of portal Hypertension at 6 & 12 months | 6 & 12 months
Improved Growth parameters at 3, 6, 12 months | 3, 6, 12 months
Reduction in Bilirubin levels at 3, 6, 12 month | 3, 6, 12 months
Reduced PELD at 3, 6, 12 months | 3, 6, 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided